CLINICAL TRIAL: NCT06788366
Title: AI-HOPE Lung Cancer: Building a Predictive Tool for Metastatic Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesca Rita Ogliari, Principal investigator, Medical doctor, IRCCS San Raffaele
Other Study IDs: AI-HOPE
Record Dates: First submitted 2024-02-29; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mono-immunotherapy: Patients with NSCLC stage IV treated with immunotherapy alone as first-line treatment
  Interventions: Drug: Immunotherapy
- Chemo-immunotherapy: Patients with NSCLC stage IV treated with chemo-immunotherapy as first-line treatment
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Immunotherapy — First-line regimen according to clinical practice
Drug: Chemotherapy — First-line regimen according to clinical practice
  Groups: Chemo-immunotherapy

SUMMARY:
The goal of our project is building a predictive response algorithm for patients with metastatic lung cancer, exploiting an artificial intelligence platform. It will collect patient information from all areas (clinical, laboratory, radiological, pathological) and analyse them, understanding connections and correlations, both at baseline and at pre-specified timepoints. It would lead to the development of a reliable and constantly evolving predictive score, able to continuously re-weight the importance of each variable as new data come in.

Since the greatest clinical need is identifying non-responders to immunotherapy and chemo-immunotherapy combination (30% of all treated patients), these two populations are defined as the starting cohorts (Cohort A, immunotherapy alone, Cohort B, chemo-immunotherapy combinations).

For each cohort, three main questions are to be answered:

Q1) Early progressors (defined as progressive disease or death within three months of treatment or at first radiological restaging) Q2) Toxicity (with a special focus on severe toxicities G≥3) Q3) Long survivors (defined as patients reaching an overall survival of at least 1.5x median overall survival in registrative trials)

The early identification of non-responders, high-risk patients (or on the other hand, long survivors) would help their healthcare planning, providing individualised follow-up strategies or prompting their inclusion in alternative treatments (eg clinical trials).

For all cohorts, first data entry will be retrospective and second data entry will be prospective (as validation set).

ELIGIBILITY:
Inclusion criteria:

* Patients with histological or cytological diagnosis of NSCLC
* Stage IV according to investigator's staging procedures (or any locally advanced tumour not feasible for local radical treatment)
* Treatment with at least 1 cycle of mono-immunotherapy or chemo-immunotherapy (as per clinical practice)
* Availability of follow-up

Exclusion criteria:

* Patients with other thoracic tumours non-NSCLC (i.e. SCLC)
* Stage other than IV or feasible for radical treatment upfront
* Treatment within clinical trials (with combination regimens different from the aforementioned combinations)
* Lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC stage IV treated with at least 1 cycle of first-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Early progressive disease | From date of enrolment until the date of first documented disease progression or death, whichever comes first, assessed within 8 to 12 weeks from first-line treatment start
  Number of patients experiencing progressive disease (PD) as best response to first-line treatment
Lung toxicity | From date of enrolment until the date of first documented immune-related pneumonitis of G3 or more, assessed up to 96 months
  Number of patients experiencing immune-related pneumonitis of G3 or more
Long survivors | At a 3-year cut-off
  Numbero of patients experiencing an overall survival (time from treatment initiation to death) longer than 3 years (1.5x median overall survival from clinical trials)

CONTACTS AND LOCATIONS:
Locations (1):
- Francesca Rita Ogliari, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT06788366/Prot_SAP_000.pdf